CLINICAL TRIAL: NCT00662259
Title: Randomized, Double-blind, Placebo-controlled Study of a Benzodiazepine vs Placebo on Functional Magnetic Resonance Imaging (fMRI) of the Brain, and on Behavioral/Clinical Measures in Patients With Generalized Anxiety Disorder
Brief Title: Drug Treatment Validation of Functional Magnetic Resonance Imaging in Generalized Anxiety Disorder
Acronym: GAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Gregory G. Brown, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WP21030
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-06

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety disorders; Generalized anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- alprazolam (Experimental): Alprazolam, an FDA-approved drug, will be administered to 24 patients with generalized anxiety disorder.
  Interventions: Drug: Alprazolam (Xanax)
- placebo (Placebo Comparator): A placebo comparator will be administered to 12 patients with generalized anxiety disorder
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alprazolam (Xanax) — Drug dose will be fixed across patients: alprazolam 0.5 mg b.i.d escalating to 1.0 mg b.i.d. The treatment duration will be approximately 28 days (4 weeks).
  Other Names: Xanax
  Arms: alprazolam
Drug: Placebo — Placebo, bid, p.o. for 28 +/- 2 days.
  Arms: placebo

SUMMARY:
The purpose of this study is to find out how an anti-anxiety drug or placebo affects the activity of your brain when you are at rest and when you are viewing emotional material, such as, emotional faces and pictures.

DETAILED DESCRIPTION:
This is an exploratory study to evaluate the usefulness of fMRI as a biomarker to measure the response to a known, FDA approved marketed anxiolytic. As such, this is not a study testing safety and efficacy of an approved medicine; it is a study to evaluate the usefulness of fMRI (a non-significant risk device procedure) to correlate the clinical/behavioral effects of a marketed anxiolytic with brain activity assessed by magnetic resonance imaging. fMRI is a more direct measure of brain function than behavior, outcomes are quantitative and objective. As such, it may be more specific, i.e., may be more sensitive to drug effects or show them earlier than clinical endpoints and enable determination of efficacy in smaller or shorter studies than those required to show effects on clinical endpoints. Finally, imaging may allow differentiation of placebo responders from true drug responders.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 - 65 years of age, inclusive
2. In good general health (as determined by medical history, physical examination, laboratory assessments and electrocardiogram (ECG)), especially no findings (including concomitant medications) that would constitute contraindications for treatment with alprazolam
3. Diagnostic and Statistical Manual-IV criteria for Generalized Anxiety Disorder (GAD) (exception: at least 3 months of symptoms)
4. Hamilton Anxiety Scale at screening >/= 20
5. Montgomery-Asberg Depression Rating Scale (MADRS) at screening < 25
6. Prior medications washout:

   * 2-week medication washout prior to randomization for most psychotropic medications
   * If prior history of fluoxetine use, this drug must have been discontinued at least 5 weeks before randomization
7. For females of non-childbearing potential: either postmenopausal for the past year (confirmed by an follicle stimulating hormone level greater than 40 mIU/mL unless the subject is receiving hormone replacement therapy), or surgically sterile (e.g., tubal ligation, hysterectomy)
8. Males and female subjects of child-bearing potential may be included if using appropriate contraceptive methods:

   * must use abstinence or two methods of contraception throughout the trial:

     * should include one primary (e.g., systemic hormonal contraception, vasectomy of the male partner) AND one secondary barrier method (e.g., latex condoms, spermicide) OR
     * a double barrier method (e.g., latex condom plus spermicide (foam, suppository, gel, cream)) may be used
9. GAD should be the clinically predominant disorder, as judged by the investigator, considering relative severity and impact on functioning

Exclusion Criteria:

1. Axis I disorder other than stated above with the exception of the following permitted comorbidities:

   * history of (within past 6 months) or current dysthymia
   * current (within past 6 months) depressive episode with MADRS at baseline < 25
   * history of major depression as long as no current depressive episode as defined above
2. Drug or alcohol dependence in the past 6 months
3. Positive urine toxicology (drugs of abuse as determined by clinician's assessment of positive urine test)
4. Active suicidal ideation (determined by clinician)
5. For females of childbearing potential: Pregnancy or intent to become pregnant or currently breastfeeding
6. Current use of beta-blockers or stimulants (e.g., Methylphenidate, d-Amphetamine, modafinil, and illicit drugs like cocaine or 3,4-methylenedioxy-N-methylamphetamine [MDMA])
7. Current regular use of antihistamines (except for inhalants which are permitted)
8. Current use of herbal medication for mood or anxiety disorders and unwillingness to discontinue use for the duration of the study
9. Current use of fluoxetine
10. Concomitant psychotropic medications including regular use of sleeping medications (also herbals)

    * occasional use of sleeping medication, with the exception of benzodiazepines, is permitted as long as it is not taken the evening prior to a visit
11. Past intolerance (including allergic) to, or clear history of non-response to the study medication
12. Current smoker (> 10 cigarettes/day); habitual caffeine consumption of more than 400 mg/d (approximately 4 cups of coffee or equivalent)
13. Body mass index > 32.5 kg/m2
14. Contraindication to magnetic resonance imaging based on a standard fMRI screening forms
15. Concurrent participation in an institutional review board (IRB) approved investigational drug trial
16. Any other reason why, per clinician, the patient should not participate in this study (to be included in this assessment are all considerations, warnings, precautions as per current FDA-approved drug label for Xanax®)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Paulus MP, Feinstein JS, Castillo G, Simmons AN, Stein MB. Dose-dependent decrease of activation in bilateral amygdala and insula by lorazepam during emotion processing. Arch Gen Psychiatry. 2005 Mar;62(3):282-8. doi: 10.1001/archpsyc.62.3.282. PMID 15753241
- [Background] Salmeron BJ, Stein EA. Pharmacological applications of magnetic resonance imaging. Psychopharmacol Bull. 2002 Winter;36(1):102-29. PMID 12397851
- [Background] Simmons A, Strigo I, Matthews SC, Paulus MP, Stein MB. Anticipation of aversive visual stimuli is associated with increased insula activation in anxiety-prone subjects. Biol Psychiatry. 2006 Aug 15;60(4):402-9. doi: 10.1016/j.biopsych.2006.04.038. PMID 16919527
- [Background] Baas JM, Grillon C, Bocker KB, Brack AA, Morgan CA 3rd, Kenemans JL, Verbaten MN. Benzodiazepines have no effect on fear-potentiated startle in humans. Psychopharmacology (Berl). 2002 May;161(3):233-47. doi: 10.1007/s00213-002-1011-8. Epub 2002 Mar 20. PMID 12021826
- [Background] Grillon C, Baas JM, Pine DS, Lissek S, Lawley M, Ellis V, Levine J. The benzodiazepine alprazolam dissociates contextual fear from cued fear in humans as assessed by fear-potentiated startle. Biol Psychiatry. 2006 Oct 1;60(7):760-6. doi: 10.1016/j.biopsych.2005.11.027. Epub 2006 Apr 21. PMID 16631127

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alprazolam | Placebo
Started | 21 | 11
Completed | 19 | 11
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alprazolam | Placebo | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.63 (14.77) | 36.27 (14.69) | 37.8 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 19 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 9 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Signal Change in Brain Activity in the Amygdala When Viewing Emotional Faces
Description: Extent of activation a brain signal when matching emotional face expressions as a percentage of the brain signal when matching geometric designs. The brain signal is the blood oxygen level dependent signal measured by functional magnetic resonance imaging.
Time Frame: 0,1,28 days
Population: 19 out of 21 participants analyzed due to 2 withdrawing from adverse events.
Measure: Mean (Standard Deviation); unit: Percent signal change in brain acitivity
Arm/Group | Alprazolam | Placebo
Number analyzed (Participants) | 19 | 11
Percent signal change in brain acitivity
  Day 0 (Baseline) | .1489 (.1529) | .1074 (.1123)
  Day 1 | .0119 (.1050) | .1404 (.0987)
  Day 28 | .1230 (.1366) | .1699 (.1058)

2. Primary Outcome: Signal Change in Brain Activity in the Insula When Anticipating the Viewing of Emotional Pictures.
Description: Extent of activation of a brain signal when anticipating the viewing of an emotional picture as a percentage of brain signal when the viewing of an emotional signal is not anticipated. The brain signal is the blood oxygen level dependent signal as measured by functional magnetic resonance imaging.
Time Frame: 0,1,28 days
Population: Nineteen of 21 alprazolam participants analyzed to two subjects withdrawing due to adverse events.
Measure: Mean (Standard Deviation); unit: Percent signal change in brain acitivity
Arm/Group | Alprazolam | Placebo
Number analyzed (Participants) | 19 | 11
Percent signal change in brain acitivity
  Day 0 (Baseline) | .0707 (.0322) | .0724 (.0522)
  Day 1 | .0458 (.0274) | .0645 (.0310)
  Day 28 | .0596 (.0426) | .0461 (.0337)

3. Secondary Outcome: Score on the Hamilton Anxiety Scale
Description: Measured participant's general anxiety; range 0 - 56; higher scores worse
Time Frame: 0, 7, 28 days
Population: Nineteen of 21 participants analyzed due to two participants withdrawing due to adverse events.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alprazolam | Placebo
Number analyzed (Participants) | 19 | 11
score on a scale
  Day 0 (Baseline) | 27.79 (5.99) | 28.00 (5.42)
  Day 7 | 13.58 (6.94) | 22.18 (6.71)
  Day 28 | 10.85 (6.01) | 20.18 (8.74)

4. Secondary Outcome: Score on the Penn State Worry Scale
Description: Measured participant's extent of worry; range 16 - 80, higher scores worse
Time Frame: 0, 7, 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alprazolam | Placebo
Number analyzed (Participants) | 19 | 11
score on a scale
  Day 0 (Baseline) | 64.74 (8.31) | 66.73 (7.76)
  Day 7 | 50.26 (10.57) | 62.45 (7.58)
  Day 28 | 48.11 (12.28) | 61.36 (10.33)

5. Other Pre Specified Outcome: Score on Quick Inventory of Depressive Symptomatology
Description: Measured the level of a participant's depression; 0 - 48; higher scores worse
Time Frame: 0, 7, 28 days
Population: Nineteen of 21 participants analyzed due to 2 participants withdrawal due to adverse events.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alprazolam | Placebo
Number analyzed (Participants) | 19 | 11
score on a scale
  Day 0 (Baseline) | 12.42 (4.90) | 12.09 (4.35)
  Day 7 | 8.05 (4.96) | 10.09 (3.83)
  Day 28 | 6.42 (3.36) | 9.09 (3.30)

ADVERSE EVENTS:
Time Frame: From day 0 (baseline) to day 28.
Arm/Group | Alprazolam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 2/21 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprazolam (N=21) | Placebo (N=11)
Drowsiness (Psychiatric disorders) | 1 (1) | 0 (0)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes